CLINICAL TRIAL: NCT05286515
Title: A Pilot Study to Test the Feasibility of a Hybrid Preoperative Physical Therapy Intervention for Patients Undergoing Total Joint Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-01331
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Total Joint Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Preoperative Physical Therapy (PT) (Experimental)
  Interventions: Other: Hybrid Peroperative PT
- Control Standard Physical Therapy (PT) (Active Comparator)
  Interventions: Other: Standard Clinical Practice PT

INTERVENTIONS:
Other: Hybrid Peroperative PT — The intervention will consist of an in-person evaluation assessing the subject's functional level, lower and upper extremities range of motion, strength and endurance. The remaining sessions will be conducted via telehealth. The program will consist of two sessions per week up to six weeks. The program will start approximately 8 to 7 weeks before the scheduled surgery date.
  Arms: Hybrid Preoperative Physical Therapy (PT)
Other: Standard Clinical Practice PT — This group will follow the protocols established by the PT facility they chose. They will finish treatment two to three weeks before the surgery date, similar to the intervention group.
  Arms: Control Standard Physical Therapy (PT)

SUMMARY:
This study aims to determine the feasibility of implementing a hybrid physical therapy intervention prior to total joint replacement surgery.

DETAILED DESCRIPTION:
Study objectives include: 1) testing the feasibility of a hybrid preoperative physical therapy intervention for physically deconditioned patients undergoing total hip and knee replacement, and 2) observing differences in post-surgical outcomes such as pain, pain interference, function and healthcare utilization, between patients who receive the intervention and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Patient is above 55 years old, indicated for primary total knee or hip replacement surgery and is deconditioned based on the surgeon's clinical judgement (i.e., Use of walker, limited or staggered gait, difficulty in sit to stand) as recorded in study log.
* Patient falls below the median score on the HOOS/KOOS JR/PROMIS physical function (<47.4, <49.8, ≤ 37 respectively and below the median score on the PROMIS Pain Interference score (≥63).
* Patient has access to technology to participate in telehealth.

Exclusion Criteria:

* Patient is not ambulatory
* Patient is scheduled for bilateral arthroplasty or revision arthroplasty.
* Patient is morbidly obese (BMI >40).
* Patient has pre-existing medical condition that is contraindicated for exercise such as unstable cardiomyopathy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference - Short Form 6b | Baseline, Month 2
  PROMIS - Pain Interference - Short Form 6b measure the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional physical, and recreational activities. Pain Interference items utilize a 7-day recall period ("the past 7 days"). PROMIS - PI - Short Form 6b consists of 6 items. Each question is scored between 1 to 5. The total score range is 6-30; the higher the score the more of the concept is being measured (more pain interference).
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference - Short Form 6b | Month 2, Month 5
  PROMIS - Pain Interference - Short Form 6b measure the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional physical, and recreational activities. Pain Interference items utilize a 7-day recall period ("the past 7 days"). PROMIS - PI - Short Form 6b consists of 6 items. Each question is scored between 1 to 5. The total score range is 6-30; the higher the score the more of the concept is being measured (more pain interference).

SECONDARY OUTCOMES:
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Intensity - Short Form 3a | Baseline, Month 2
  PROMIS - Pain Intensity - Short Form 3a consists of 3 questions -- participants report on the intensity of pain experienced in the past 7 days. Each question is scored between 1 (had no pain) to 5 (very severe). The total score range is 3-15; the higher the score, the more intense the pain.
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Intensity - Short Form 3a | Month 2, Month 5
  PROMIS - Pain Intensity - Short Form 3a consists of 3 questions -- participants report on the intensity of pain experienced in the past 7 days. Each question is scored between 1 (had no pain) to 5 (very severe). The total score range is 3-15; the higher the score, the more intense the pain.
Change in Score on Patient-Reported Outcomes Measurement Information System - Physical Function - 10 (PROMIS-PF-10) | Baseline, Month 2
  PROMIS-PF-10 consists of 10 items. Item-levels are scored numerically for an individual's response to each question. The total score range is 10-100; higher scores mean more of a concept being measured (e.g., more fatigue).
Change in Score on Patient-Reported Outcomes Measurement Information System - Physical Function - 10 (PROMIS-PF-10) | Month 2, Month 5
  PROMIS-PF-10 consists of 10 items. Item-levels are scored numerically for an individual's response to each question. The total score range is 10-100; higher scores mean more of a concept being measured (e.g., more fatigue).
Change in Hip Disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS, JR) | Baseline, Month 2
  HOOS, JR contains 6 items from the original HOOS survey. Items are coded from 0 to 4, none to extreme, respectively. HOOS, JR is scored by summing the raw response (range 0-24) and then converting it to an interval score. The interval score ranges from 0-100, where 0 represents total hip disability and 100 represents perfect hip health.
Change in Hip Disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS, JR) | Month 2, Month 5
  HOOS, JR contains 6 items from the original HOOS survey. Items are coded from 0 to 4, none to extreme, respectively. HOOS, JR is scored by summing the raw response (range 0-24) and then converting it to an interval score. The interval score ranges from 0-100, where 0 represents total hip disability and 100 represents perfect hip health.
Change in Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Baseline, Month 2
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Change in Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | Month 2, Month 5
  KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Average Number of Physical Therapy Sessions Since Enrollment in the Study | Month 2
  Self-reported
Average Number of Times Per Week Participants Had Physical Therapy | Month 2
  Self-reported
Number of Readmissions | Month 5
  Self-reported hospital readmission for any reason including revision surgery ED visits

OTHER OUTCOMES:
Baseline Score on General Anxiety Disorder Screener (GAD-7) | Baseline
  GAD-7 consists of 7 problems. Participants report how often they have been bothered by the 7 problems over the last 2 weeks on a Likert Scale from 0 (not at all) to 3 (nearly every day). The total score range is 0-21; the higher the score, the more severe the anxiety. 0-4=minimal anxiety, 5-9=mild, 10-14=moderate, 15-21=severe anxiety.
Baseline Score on Center for Epidemiologic Studies Depression Scale Revised-10 (CESD-R-10) | Baseline
  CED-R-10 is a self-report measure of depression consisting of 10 items. The total score is calculated by finding the sum of the items with a range of 0-30. The higher the score, the greater the depression. Any score equal to or above 10 is considered depressed.
Score on Measuring Patient Satisfaction (MRPS) Scale | Month 2
  MRPS consists of 8 items. The rating scale of each item goes from 1 to 5 where 1 is 'strongly disagree' and 5 is 'strongly agree.' The score is calculated as the sum of the item scores with a total score range of 8-40; where a higher score represents higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Campello, PT, PhD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Occupational & Industrial Orthopaedic Center (OIOC), New York, New York
  - NYU Langone Orthopedic Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Marco.Campello@nyulangone.org to gain access, data requestors will need to sign a data access agreement.